CLINICAL TRIAL: NCT05180175
Title: The Nordic IBD Treatment Strategy Trial- a Randomised Controlled Trial of Access to a Protein Profile
Brief Title: The Nordic IBD Treatment Strategy Trial
Acronym: NORDTREAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NT-2020
Record Dates: First submitted 2021-12-17; First posted 2022-01-06 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to protein profile (Experimental)
  Interventions: Drug: Top down treatment if patient at high risk
- No access to protein profile (No Intervention)

INTERVENTIONS:
Drug: Top down treatment if patient at high risk — Patients with an increased risk of poor disease course (as defined by a serum protein signature at diagnosis), will be treated with a top down treatment strategy.
  Arms: Access to protein profile

SUMMARY:
Purpose:

To demonstrate that personalised therapy can be delivered to patients with IBD, by treating patients with an increased risk of poor disease course, defined by a serum protein signature at diagnosis, with a top-down treatment, and that this treatment strategy improves clinical outcomes.

Objectives:

Primary objective: To assess if a top-down treatment can improve treatment outcomes in IBD patients with a high risk of poor disease course, defined by a serum protein signature at diagnosis.

Secondary objective: To assess if a top-down treatment can improve quality of life and health resource allocation in IBD patients with a high risk of poor disease course, defined by a serum protein signature at diagnosis.

Study design:

A multi-centre, biomarker-stratified open-label controlled trial, where newly diagnosed IBD patients are randomised (1:1) to a group with access to the protein signature or a group without access to the protein signature. Study subjects within the protein signature arm who display a high-risk protein profile, will be treated according to a top-down treatment algorithm (anti-TNF agent with/without an immunomodulatory) and subjects without access to the protein signature will be treated according to current clinical practice.

Study population:

Newly diagnosed IBD patients.

Number of subjects: 300

Primary variables:

Composite of both corticosteroid-free clinical remission and endoscopic remission at Week 52, defined as below. Surgery because of IBD during follow-up will be defined as treatment failure.

Ulcerative colitis;

* Clinical remission per patient reported Mayo: A stool frequency subscore (SFS) ≤ 1, and not greater than baseline, and a rectal bleeding subscore (RBS) of 0.
* Endoscopic remission: An endoscopic Mayo subscore of 0 (OR in patients without endoscopy at week 52, normalization of f-Calprotectin, defined as < 250μg/g

Crohn's disease;

* Clinical remission: An average daily Stool Frequency (SF) ≤ 2.8 and not worse than Baseline AND average daily Abdominal Pain (AP) score ≤ 1 and not worse than Baseline.
* Endoscopic remission: SES-CD≤2 (OR in patients without endoscopy at week 52, normalization of f-Calprotectin, defined as < 250μg/g.

ELIGIBILITY:
Inclusion Criteria:

* UC or CD diagnosed within < 4 weeks using standard endoscopic, histologic or radiological criteria (ECCO Criteria). Histology report may not be available at baseline.
* Naïve to immunomodulators, biologics and small molecules, i.e. JAK-inhibitors
* Aged 18-70 years old.
* Is considered eligible according to tuberculosis (TB) screening criteria.
* Written informed consent to participate in the study

Exclusion Criteria:

* A previous known diagnosis of Crohn's disease, ulcerative colitis or IBD-U, since >6 weeks before baseline
* Unable to provide informed consent
* Unable to comply with protocol requirements (e.g. for reasons including alcohol and/or recreational drug abuse)
* Ongoing sepsis
* Acute obstructive symptoms AND evidence of a fixed stricture on radiology or colonoscopy, which suggest that the patient is in need of surgery over the following year. N.B. patients with modest degrees of stricturing on imaging but no obstructive symptoms may be included according to clinician judgement
* Contra-indications to trial medications including a history of hepatitis B or C, tuberculosis, Cardiac failure, NYHA III-IV or hypersensitivity. Hypersenstitivity to a thiopurine agent should alert the prescriber to probable hypersensitivity to other thiopurines.
* History of malignancy
* Pregnancy at baseline
* Other serious medical or psychiatric illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Clinical and endoscopic remission | Week 52
  Composite of proportion of subjects with both corticosteroid-free clinical remission and endoscopic remission at Week 52. Surgery because of IBD during follow-up will be defined as treatment failure.

SECONDARY OUTCOMES:
Clinical/Endoscopy remission and response | Week 52
  1. Proportion of subjects with clinical remission at 52 weeks
  2. Proportion of subjects with endoscopic remission at 52 weeks
  3. Proportion of subjects with clinical response
  4. Proportion of subjects with endoscopic response
  5. The proportion of patients with drug-related adverse events

CONTACTS AND LOCATIONS:
Locations (15):
- Denmark (3):
  - Hospital Sønderjylland, Aabenraa
  - Odense University Hospital, Odense
  - OUH Svendborg Hospital, Svendborg
- Landspitali, Reykjavik, Iceland
- Norway (5):
  - Vestre Viken HF, Drammen
  - Østfold Kalnes, Grålum
  - Oslo Universitetssykehus, Oslo
  - Sykehuset i Telemark, Skien
  - Sykehuset i Vestfold, Tønsberg
- Sweden (6):
  - Höglandssjukhuset Eksjö, Eksjö, Region Jönköpings Län
  - Karolinska Universitetssjukhuset, Stockholm, Region Stockholm
  - Akademiska Sjukhuet Uppsala, Uppsala, Region Uppsala
  - Universitetssjukhuset i Linköping, Linköping, Region Östergötland
  - Ersta sjukhus, Stockholm, Stockholm County
  - Universitetssjukhuset Örebro, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rejler M, Fuchtbauer JD, Daviethsdottir LG, Fejrskov A, Soderholm JD, Christensen R, Andersen V, Repsilber D, Kjeldsen J, Hoivik M, Halfvarson J. Nordic inflammatory bowel disease treatment strategy trial: protocol for the NORDTREAT randomised controlled biomarker-strategy trial. BMJ Open. 2024 Jul 31;14(7):e083163. doi: 10.1136/bmjopen-2023-083163. PMID 39089718